CLINICAL TRIAL: NCT07160283
Title: The Efficacy and Safety of Trilaciclib in Bone Marrow Protection Before Chemotherapy for Advanced Bile Duct Cancer and Pancreatic Cancer
Status: Not yet recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: The Second Affiliated Hospital of Shandong First Medical University (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: MT-008
Record Dates: First submitted 2025-08-16; First posted 2025-09-08 (Actual); Last update posted 2025-09-08 (Actual); Status verified 2025-08

CONDITIONS: Biliary Tract Neoplasms; Pancreatic Neoplasms
MeSH Terms: conditions — Biliary Tract Neoplasms; Pancreatic Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Trilaciclib combined with chemotherapy for the treatment of advanced cholangiocarcinoma and pancreat (Experimental): Trilaciclib: 240 mg/m², administered via intravenous infusion over 30 minutes, completed within 4 hours prior to chemotherapy on the same day.
  Chemotherapy Agents: Investigators will select chemotherapy regimens based on individual patient status. Regimens must be single-day protocols (including but not limited to gemcitabine, nab-paclitaxel, etc.), with dosing and administration per prescribing information.
  Subjects receiving concomitant immunotherapy or targeted therapy in addition to chemotherapy are eligible for enrollment.
  Interventions: Drug: Bile duct cancer cohort; Drug: Pancreatic cancer cohort

INTERVENTIONS:
Drug: Bile duct cancer cohort — Trilaciclib: 240 mg/m², administered via intravenous infusion over 30 minutes, completed within 4 hours prior to chemotherapy on the same day.
  Chemotherapy Agents: Investigators will select chemotherapy regimens based on individual patient status. Regimens must be single-day protocols (including but not limited to gemcitabine, nab-paclitaxel, etc.), with dosing and administration per prescribing information.
  Subjects receiving concomitant immunotherapy or targeted therapy in addition to chemotherapy are eligible for enrollment.
Drug: Pancreatic cancer cohort — rilaciclib: 240 mg/m², administered via intravenous infusion over 30 minutes, completed within 4 hours prior to chemotherapy on the same day.
  Chemotherapy Agents: Investigators will select chemotherapy regimens based on individual patient status. Regimens must be single-day protocols (including but not limited to gemcitabine, nab-paclitaxel, etc.), with dosing and administration per prescribing information.
  Subjects receiving concomitant immunotherapy or targeted therapy in addition to chemotherapy are eligible for enrollment.

SUMMARY:
Evaluate the efficacy and safety of Trilaciclib for myeloprotection prior to chemotherapy in advanced cholangiocarcinoma or pancreatic cancer.

ELIGIBILITY:
Inclusion Criteria:

1. Age >18 years, male or female.
2. Pathologically confirmed diagnosis of cholangiocarcinoma or pancreatic cancer requiring chemotherapy-based treatment.
3. ECOG performance status ≥0 (or 1), anticipated survival ≥3 months, and ability to complete ≥3 months of follow-up.
4. No clinically significant abnormalities in complete blood count, hepatic/renal function, cardiac enzymes, or electrocardiogram (ECG).
5. Voluntary participation with good compliance and willingness to undergo safety and survival follow-up.
6. Signed written informed consent form prior to enrollment.

Exclusion Criteria:

1. History of myeloid leukemia, myelodysplastic syndrome, or concurrent sickle cell disease.
2. Symptomatic CNS metastases and/or leptomeningeal disease requiring immediate radiotherapy or steroid therapy.
3. Major surgery or radiotherapy within 4 weeks prior to the first dose of study drug.
4. History of interstitial lung disease, slowly progressive dyspnea with dry cough, sarcoidosis, silicosis, idiopathic pulmonary fibrosis, pulmonary hypersensitivity pneumonitis, multiple allergies, or peripheral arterial disease.
5. Concurrent requirement for radiotherapy.
6. Known hypersensitivity to any component of the study drug formulation.
7. Pregnancy or lactation.
8. Any other condition deemed by the investigator to compromise patient safety or study validity.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 96 (Estimated)
Dates: Start 2025-09-01 (Estimated); Primary Completion 2027-09-01 (Estimated); Study Completion 2028-09-01 (Estimated)

PRIMARY OUTCOMES:
Incidence of Grade ≥3 Chemotherapy-Induced Neutropenia (CIN) During Chemotherapy Cycles | through study completion, an average of 1 year

SECONDARY OUTCOMES:
The incidence of grade ≥ 3 thrombocytopenia | through study completion, an average of 1 year
The incidence of FN | through study completion, an average of 1 year

OTHER OUTCOMES:
OS | 2 years
  Throughout the Entire Chemotherapy Course
PFS | 1 year
  The length of time during and after the treatment of a disease, such as cancer, that a patient lives with the disease but it does not get worse

CONTACTS AND LOCATIONS:
Overall Officials: yan hai Liu, Principal Investigator — The Second Affiliated Hospital of Shandong First Medical University

IPD SHARING:
Plan to Share IPD: No